CLINICAL TRIAL: NCT06701617
Title: The Effectiveness of In-person and Telehealth Visual Rehabilitation for Children With Low Vision
Brief Title: In-person and Telehealth Visual Rehabilitation for Children With Low Vision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202306050RINC
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Visual Rehabilitation; Oddball Design; Cerebral Visual Impairment; Passive Visual Stimulation; Perceptual Learning
Keywords: visual rehabilitation; visual stimulation; perceptual learning
MeSH Terms: conditions — Blindness, Cortical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Visual rehabilitation group (Experimental): This study includes two distinct groups: one comprising individuals with non-severe visual impairment and the other consisting of individuals with severe or profound visual impairment. The severe/profound visual impairment group receives passive visual stimulation, while the non-severe visual impairment group undergoes visual stimulation using a checkerboard pattern. The latter approach incorporates perceptual learning theories, emphasizing attentional modulation and leveraging the oddball design concept to enhance visual processing and rehabilitation outcomes.
  Interventions: Behavioral: restorative visual rehabitation
- Usual care group (No Intervention): Usual care includes physical games and teaching methods that utilize auditory and tactile senses to compensate for vision.

INTERVENTIONS:
Behavioral: restorative visual rehabitation — black-and-white checkerboard patterns, visual stimulation program, restorative visual rehabitation
  Arms: Visual rehabilitation group

SUMMARY:
Restorative visual rehabilitation is frequently used to enhance the visual development and function of children with low vision. An important strategy within this field is visual stimulation, which is particularly used for infants and toddlers with low vision, as well as for children who have both developmental disabilities and low vision.This study has two primary objectives.The first objective is to examine the effect of using intensive, specific, and flickering black-and-white checkerboard patterns to enhance visual function in children with mild to moderate low vision. The second objective is to develop a visual stimulation program tailored for children with severe or profound multiple disabilities and visual impairments, and to evaluate its effectiveness.

DETAILED DESCRIPTION:
Investigators will recruit 200 children with various types and severities of visual disorders. Additionally, investigators will collect eye movement assessment data using an eye-tracking system from 30 typically developing infants under two years old to validate the oculomotor assessment newly designed for this study. For this component, the reliability of our oculomotor assessment will be validated through test-retest reliability in both typically developing children and children with multiple disabilities and visual impairments who are enrolled in visual rehabilitation.

The intervention programs include two types:

1. One program provides extensive passive visual stimulation, incorporating attentional modulation during the process to facilitate training. Passive visual stimulation is delivered continuously using appropriate visual materials tailored to the participants' visual abilities, such as illuminated toys or high-contrast patterns. These stimuli are positioned around infants or children, or repeatedly presented by caregivers. This approach allows young children or those with lower cognitive abilities and visual impairments to receive visual stimulation even without active participation. Through this passive intervention model, visual function can be improved.

   Although this model is flexible and suitable for infants or children with low compliance, it poses challenges in quantifying the amount of visual training provided. This limitation affects the ability to verify the efficacy of interventions in clinical trials.

   This version incorporates technical terms and ensures clarity for academic or clinical documentation, while emphasizing the model's flexibility and its limitations.
2. Another program provide checkerboard pattern, a fundamental visual element processed by the early vision system, is used widely in vision science research, visual function assessment, and training. This program incorporates perceptual learning theories that emphasize attentional modulation and the oddball design concept. Salient oddball patterns appear randomly within the ongoing checkerboard reversal stimuli. Participants are required to press a special button when these patterns appear, with engaging auditory feedback provided to reinforce correct responses. This design aims to sustain the visual attention of visually impaired infants and children on the checkerboard reversal patterns for longer durations. Neurologically, the program strengthens top-down modulation mechanisms in the brain through random salient stimuli, enhancing bottom-up processing of early visual information.

Researchers adjusted square sizes through trial-and-error and clinical experience, often enlarging the squares to engage the children effectively. However, this strategy may not fully accommodate children with low vision combined with developmental disabilities. Behavioral observations suggest that integrating sVEP to identify occipital response thresholds and utilizing eye-tracking systems could refine square size adjustments and improve intervention strategies and outcome evaluations.

Additionally, this program may not be suitable for children with severe or profound low vision. The need for quick physical or verbal responses to transient oddball stimuli and the requirement to recognize checkerboard patterns demand a certain level of visual acuity and sustained attention. These factors pose challenges for children with severe multiple disabilities (MDVI), who often require longer response times, have shorter attention spans, and struggle with repetitive tasks. Despite these challenges, MDVI children exhibit visual plasticity, making visual stimulation interventions valuable. Developing alternative visual stimulation programs tailored to the needs of children with severe or profound MDVI is essential for maximizing their potential benefits.

ELIGIBILITY:
Passive visual stimulation group

Inclusion Criteria:

1. Children aged less than or equal to 12 years old.
2. The causes of visual disorder in children are unlimited.
3. The acuity of children's better eye ranges between hand move and 0.2.
4. Children with multiple disabilities and visual disorders typically exhibit developmental levels ranging from moderate to severe or below.
5. The parents of these children exhibit a positive attitude and are willing to cooperate with visual learning programs.
6. Infants under 1 year old with low vision without other developmental issues , under or equal to moderate developmental issues.

Exclusion Criteria:

1. Significant refractive errors that affect acuity but are unable to cooperate with wearing corrective glasses in two training sessions.
2. Requires patching for monocular vision rehabilitation but is unable to cooperate with patching in two training sessions.
3. The individual is unable to adapt to the training environment and cooperate with visual learning in two sessions due to unstable emotions or difficulty adapting to the environment.

Perceptual learning group Inclusion Criteria

1. Children aged less than or equal to 12 years old.
2. No restrictions on the causes of visual impairment in children.
3. Best-corrected visual acuity (BCVA) in the better eye is equal to or better than 0.02.
4. If children have additional developmental issues, their disability severity should primarily be mild or moderate.
5. The primary caregiver demonstrates a positive attitude and is willing to cooperate with the visual training program.
6. The child is capable of completing calibration with an eye-tracking device. Exclusion Criteria

(1)Significant refractive errors that severely affect vision, where the child cannot adapt to wearing corrective glasses within two training sessions.

(2)Requires occlusion therapy for monocular visual rehabilitation but cannot cooperate with occlusion within two training sessions.

(3)Inability to adapt to the training environment or cooperate with visual training due to emotional instability or difficulty adjusting within two training sessions.

(4)Unstable physiological conditions (e.g., epilepsy, sleep disturbances) that prevent consistent participation in visual training.

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-06-14 (Estimated)

PRIMARY OUTCOMES:
Visual Function Battery for Children with Special Needs | From enrollment to one year after the end of treatment
  Visual Function Battery for Children with Special Needs (VFB-CSN) is typically conducted by occupational therapists with experience in visual rehabilitation. It is a scale used to evaluate the visual function of children with special needs. It assesses eight aspects: visual reflection, eyeball asymmetry, visual acuity, contrast sensitivity, visual field, eye movements, color and shape perception, and visual attention. The scale includes 27 questions and combines standardized tests with functional assessment methods. The functional assessment method can be applied to cases that cannot cooperate with standardized tests. Children with varying degrees of visual impairment, ranging from light perception to identifiable visual targets, can be assessed using the VFB-CSN alone. The assessment scale has a maximum score of 60 and a minimum score of 0, with higher scores indicating better performance.
Functional Vision Questionnaire | From enrollment to one year after the end of treatment
  This questionnaire is completed by the primary caregiver. It is designed for children with severe central nervous system disorders, such as children with cerebral palsy, to evaluate their visual performance under different brightness conditions and during daily activities. The scale consists of 28 questions, with a maximum score of 140 and a minimum score of 28. Higher scores indicate better performance.
Eye Movement Assessment Behavioral Scale for Children | From enrollment to one year after the end of treatment
  The scoring is conducted by occupational therapists with experience in visual rehabilitation, based on their observation of the child's performance. This assessment employs an eye tracker and PowerPoint to create an eye movement assessment program before and after rehabilitation. It evaluates children's abilities in fixation, tracking, and saccadic movements in response to visual stimuli of varying sizes, contrasts, directions, speeds, and positions. The assessment scale has a maximum score of 64 and a minimum score of 8, with higher scores indicating better performance.
Near Detection Scale | From enrollment to one year after the end of treatment
  Near Detection Scale (NDS) is performed by clinicians specializing in visual issues among children with special needs to quickly assess the detection acuity of children with severe and profound visual impairment. NDS is an 18-point scale, with 0 representing no light perception and 18 representing the ability to see 0.1 cm objects on a dark green background at a viewing distance of 30 cm. Higher scores indicate better visual acuity.

SECONDARY OUTCOMES:
Three-Day Daily of Children's Daily Visual Performance | From enrollment to one year after the end of treatment
  This record is completed by the primary caregiver to document the child's visual behavior at home. The recording is conducted both before and after training to simultaneously capture the child's training activities and response status at home.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Occupational Therapy, College of Medicine, National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No